CLINICAL TRIAL: NCT06995326
Title: A Phase 1, Randomized, Double-blind, Placebo-controlled Single Ascending Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Subcutaneously Administered SGB-3383 in Healthy Volunteers
Brief Title: A Study of SGB-3383 in Healthy Subjects
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Suzhou Sanegene Bio Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SGB-3383-002
Record Dates: First submitted 2025-05-20; First posted 2025-05-29 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-05

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SGB-3383 (Experimental): SGB-3383 for sc injection
  Interventions: Drug: SGB-3383
- SGB-3383-Matching placebo (Placebo Comparator): Normal saline (0.9% NaCl) matching volume of SGB-3383 doses will be administered
  Interventions: Drug: SGB-3383-Matching placebo

INTERVENTIONS:
Drug: SGB-3383 — SGB-3383 for sc injection, single dose
  Arms: SGB-3383
Drug: SGB-3383-Matching placebo — SC injection, single dose
  Arms: SGB-3383-Matching placebo

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, pharmacokinetic (PK), and pharmacodynamic (PD) effects of SGB-3383 in healthy subjects. The study will be designed as a single ascending dose (SAD) phase, utilizing a double-blind, placebo-controlled approach.

ELIGIBILITY:
Inclusion Criteria:

* Weight ≥ 45.0 kg (female) or ≥ 50.0 kg (male), and Body Mass Index (BMI) within the range of 18.0 to 28.0 kg/m², inclusive
* Physical examination, vital signs, 12-lead electrocardiogram, and laboratory tests be normal or slightly abnormal but not clinically significant according to investigator's judgement.
* Participants must agree to use adequate contraception from signing the informed consent until 3 months after completion of the follow-up visit.
* Willing to comply with the protocol required visit schedule and visit requirements and provide written informed consent.

Exclusion Criteria:

* A history of or a current surgical or medical condition that, in the opinion of the Investigator, may put the subject at significant risk (according to Investigator's judgment) or interfere with the subject's participation in the clinical study.
* History of meningococcal infection, or subjects from occupations or living environment at risk of Neisseria meningitidis exposure.
* Positive result of hepatitis B surface antigen (HBsAg), hepatitis C virus antibody (HCV Ab), human immunodeficiency virus (HIV) antibody, or syphilis at screening.
* Alanine aminotransferase (ALT), total bilirubin (TBIL), aspartate aminotransferase (AST)> 1.5 × ULN, and deemed clinically significant by the Investigators
* QTcF values > 450 ms for male, and > 470 ms for female

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 37 (Estimated)
Dates: Start 2025-06 (Estimated); Primary Completion 2026-08 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events (AEs) | up to approximately 12 months

SECONDARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) of SGB-3383 | Up to Day 3
Area Under the Concentration-time Curve (AUC) of SGB-3383 | Up to Day 3